CLINICAL TRIAL: NCT06921941
Title: A Phase 1, Open-Label, Two-Part Study to Evaluate the Effect of a Single Oral Dose of Bemnifosbuvir/Ruzasvir Fixed Dose Combination on the Pharmacokinetics of Digoxin and Rosuvastatin in Healthy Subjects
Brief Title: Drug-drug Interaction Study of Bemnifosbuvir/Ruzasvir (BEM/RZR) and Digoxin and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-009
Record Dates: First submitted 2025-03-27; First posted 2025-04-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Digoxin vs Digoxin + BEM/RZR vs Digoxin + 2h BEM/RZR (Experimental)
  Interventions: Drug: Digoxin vs Digoxin + BEM/RZR vs Digoxin + 2h BEM/RZR
- Rosuvastatin vs Rosuvastatin + BEM/RZR vs Rosuvastatin + 2h BEM/RZR (Experimental)
  Interventions: Drug: Rosuvastatin vs Rosuvastatin + BEM/RZR vs Rosuvastatin + 2h BEM/RZR

INTERVENTIONS:
Drug: Digoxin vs Digoxin + BEM/RZR vs Digoxin + 2h BEM/RZR — Treatment-A (Digoxin): A single dose of digoxin will be administered under fasting conditions.
  Treatment-B (Digoxin + BEM/RZR): A single dose of digoxin will be co-administered a single dose of BEM/RZR under fasting conditions.
  Treatment-C (Digoxin + 2h BEM/RZR): A single dose of digoxin will be administered under fasting conditions. Then, a single dose of BEM/RZR will be administered approximately 2 hours later under fasting conditions.
  Other Names: AT-527 (BEM) and AT-038 (RZR)
  Arms: Digoxin vs Digoxin + BEM/RZR vs Digoxin + 2h BEM/RZR
Drug: Rosuvastatin vs Rosuvastatin + BEM/RZR vs Rosuvastatin + 2h BEM/RZR — Treatment-D (rosuvastatin): A single dose of rosuvastatin will be administered under fasting conditions.
  Treatment-E (rosuvastatin + BEM/RZR): A single dose of rosuvastatin will be co-administered with a single dose BEM/RZR under fasting conditions.
  Treatment-F (rosuvastatin + 2h BEM/RZR): A single dose of rosuvastatin will be administered under fasting conditions. Then, a single dose BEM/RZR will be administered approximately 2 hours later under fasting conditions.
  Other Names: AT-527 (BEM) and AT-038 (RZR)
  Arms: Rosuvastatin vs Rosuvastatin + BEM/RZR vs Rosuvastatin + 2h BEM/RZR

SUMMARY:
Drug-drug interaction study between Bemnifosbuvir/Ruzasvir and Digoxin or Rosuvastatin

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug.
* Minimum body weight of 50 kg and body mass index (BMI) of 18-30 kg/m2.
* Willing to comply with the study requirements and to provide written informed consent.

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2.
* Abuse of alcohol or drugs.
* Use of other investigational drugs within 28 days of dosing.
* Concomitant use of prescription medications, or systemic over-the-counter medications.
* Other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
PK of Digoxin and Rosuvastatin (Cmax) | Digoxin: Days 1,15, 29; Rosuvastatin: Days 1, 8, 15
PK of Digoxin and Rosuvastatin (AUC) | Digoxin: Days 1,15, 29; Rosuvastatin: Days 1, 8, 15

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Québec, Montreal, Canada